CLINICAL TRIAL: NCT02827877
Title: Use of 64Cu-DOTA-Trastuzumab PET Imaging and Molecular Markers for Prediction of Response to Trastuzumab and Pertuzum-Based Neoadjuvant Therapy
Brief Title: Cu64-DOTA-trastuzumab PET and Markers Predicting Response to Neoadjuvant Trastuzumab + Pertuzum in HER2+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16079; FWA 00000692 (Registry Identifier: Federal-wide Assurance Number)
Record Dates: First submitted 2016-04-26; First posted 2016-07-11 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: HER2 Positive Breast Carcinoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 64Cu-DOTA-trastuzumab; pertuzumab; 2C4 antibody; Magnetic Resonance Spectroscopy; Trastuzumab; PF-05280014

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trastuzumab, copper Cu 64-DOTA-trastuzumab PET) (Experimental): Patients receive trastuzumab IV over 15 minutes immediately before receiving copper Cu 64-DOTA-trastuzumab IV on day 0. Patients undergo PET scans at 18-24 and 42-48 hours, on day 1 and day 2. Within 4 days after completion of PET scans, patients receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks and pertuzumab IV over 30-60 minutes. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after 6 cycles of trastuzumab and pertuzumab.
  Interventions: Radiation: Copper Cu 64-DOTA-Trastuzumab; Other: Laboratory Biomarker Analysis; Biological: Pertuzumab; Procedure: Positron Emission Tomography; Procedure: Therapeutic Conventional Surgery; Biological: Trastuzumab

INTERVENTIONS:
Radiation: Copper Cu 64-DOTA-Trastuzumab — Given IV
  Other Names: 64Cu-DOTA-Trastuzumab
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; MoAb 2C4; Monoclonal Antibody 2C4; Perjeta; rhuMAb2C4; RO4368451
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: PET Scan
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014

SUMMARY:
This phase II trial studies how well copper Cu64-DOTA-trastuzumab positron emission tomography (PET) works in predicting response to treatment with trastuzumab and pertuzumab before surgery in patients with human epidermal growth factor receptor 2 (HER2) positive breast cancer that has spread from where it started to nearby tissue or lymph nodes. Diagnostic procedures, such as copper Cu 64 DOTA-trastuzumab PET, may help predict a patient's response to trastuzumab and pertuzumab before surgery in patients with locally advanced HER2 positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the standardized uptake value maximum (SUVmax) in patients with previously untreated HER2+ breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate if the uptake of copper 64 Cu-64-DOTA-trastuzumab, a proposed indicator of responsiveness to HER2-directed therapy, correlates with serpin peptidase inhibitor alpha-1 antiproteinase, antitrypsin, member 1 gene (SERPINA1) expression, which has been shown to be associated with estrogen receptor positive (ER+)/ HER2+ patient survival, both in the HER2+/ER+ patients and in all patients.

II. To compare uptake of copper Cu 64-DOTA-trastuzumab in the patients with complete pathologic response (pCR) versus (vs) non-pCR patients.

OUTLINE:

Patients receive trastuzumab intravenously (IV) over 15 minutes immediately before receiving copper Cu 64-DOTA-trastuzumab IV on day 0. Patients undergo PET scans at 18-24 and 42-48 hours, on day 1 and 2. Within 4 days after completion of PET scans, patients then receive trastuzumab IV over 30-90 minutes weekly or every 3 weeks and pertuzumab IV over 30-60 minutes. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo surgery after 6 cycles of trastuzumab and pertuzumab.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be women who have histological confirmation of HER2 positive breast cancer
* The primary tumor must be >= 2.0cm in size and/or have biopsy proven axillary nodes that are >= 2.0cm in size by mammography, ultrasound, or magnetic resonance imaging (MRI)
* The current cancer must over express HER2 as determined by immunohistochemistry (IHC) and/or fluorescence in situ hybridization (FISH)
* Patients may not have received prior HER2 directed therapies
* Participants must have normal cardiac ejection fraction (per label, as defined as institutional normal)
* Planned neoadjuvant therapy with six cycles of combined pertuzumab, trastuzumab and chemotherapy
* Ability to provide informed consent
* Negative Serum Pregnancy test

Exclusion Criteria:

* Participants who are not considered candidates for pertuzumab + trastuzumab + chemotherapy
* Concurrent malignancy other than non-melanoma skin cancer
* Patients must not have known metastatic disease
* Patients must not have received prior treatment for the current breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2026-09-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET)
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 54.9 [30.1 to 61.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian; Non-Hispanic or Latino | 4
  Race/Ethnicity: Black; Non-Hispanic or Latino | 2
  Race/Ethnicity: Caucasian; Hispanic or Latino | 8
  Race/Ethnicity: Caucasian; Non-Hispanic or Latino | 3
  Race/Ethnicity: Not Disclosed; Hispanic or Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response to Neoadjuvant Chemotherapy Determined at Surgery (Lumpectomy or Mastectomy).
Description: The response assessment is performed at the time of definitive surgery. Patients' disease will be staged in the conventional manner according to the AJCC. The primary endpoint is complete pathologic response defined as no evidence of residual invasive cancer in either the breast or regional lymph nodes.
Time Frame: Up to 1 year
Population: protocol patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 18
Participants
  Response | 14
  Non-response | 4

2. Other Pre Specified Outcome: SUV Measurement by 64Cu-DOTA Trastuzumab PET
Description: First Scan SUV Maximum, measurement by 64Cu-DOTA trastuzumab PET SUV is "Standard Uptake Value". SUV = tumor activity concentration x patient body weight/injected activity decay-corrected to time of scan.
Time Frame: Baseline
Population: protocol patients
Measure: Median (Full Range); unit: SUV
Arm/Group | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET)
Number analyzed (Participants) | 18
SUV | 6.6 [3.5 to 16.2]

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years.
Description: Adverse events were collected for all 18 patients.
Arm/Group | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET) (N=18)
acute hordeola of the right upper eyelid (Eye disorders) | 1
bacteriemia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trastuzumab, Copper Cu 64-DOTA-trastuzumab PET) (N=18)
10002272-Anemia (Blood and lymphatic system disorders) | 10
10040741-Sinus bradycardia (Cardiac disorders) | 1
10040752-Sinus tachycardia (Cardiac disorders) | 3
10043882-Tinnitus (Ear and labyrinth disorders) | 1
10047848-Watering eyes (Eye disorders) | 1
acute hordeola of the right upper eyelid (Eye disorders) | 1
twitching in L eye (Eye disorders) | 1
10000081-Abdominal pain (Gastrointestinal disorders) | 2
10005265-Bloating (Gastrointestinal disorders) | 1
10010774-Constipation (Gastrointestinal disorders) | 7
10012727-Diarrhea (Gastrointestinal disorders) | 14
10028130-Mucositis oral (Gastrointestinal disorders) | 5
10028813-Nausea (Gastrointestinal disorders) | 14
10047700-Vomiting (Gastrointestinal disorders) | 4
10066874-Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
dry heaving (Gastrointestinal disorders) | 1
pain - R side near the waist (Gastrointestinal disorders) | 1
rectal pressure (Gastrointestinal disorders) | 1
worsening acid reflux (Gastrointestinal disorders) | 1
10008531-Chills (General disorders) | 3
10016256-Fatigue (General disorders) | 13
10016558-Fever (General disorders) | 6
10016791-Flu like symptoms (General disorders) | 2
10033371-Pain (General disorders) | 1
10050068-Edema limbs (General disorders) | 2
10051792-Infusion related reaction (General disorders) | 2
10062466-Localized edema (General disorders) | 1
10046571-Urinary tract infection (Infections and infestations) | 1
10069138-Papulopustular rash (Infections and infestations) | 3
10006504-Bruising (Injury, poisoning and procedural complications) | 2
10001551-Alanine aminotransferase increased (Investigations) | 5
10001675-Alkaline phosphatase increased (Investigations) | 5
10003481-Aspartate aminotransferase increased (Investigations) | 4
10011368-Creatinine increased (Investigations) | 1
10025256-Lymphocyte count decreased (Investigations) | 5
10029366-Neutrophil count decreased (Investigations) | 2
10035528-Platelet count decreased (Investigations) | 3
10047900-Weight loss (Investigations) | 2
10049182-White blood cell decreased (Investigations) | 3
10002646-Anorexia (Metabolism and nutrition disorders) | 3
10020587-Hypercalcemia (Metabolism and nutrition disorders) | 1
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 1
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 3
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 2
10021018-Hypokalemia (Metabolism and nutrition disorders) | 4
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 1
10021038-Hyponatremia (Metabolism and nutrition disorders) | 5
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 2
increased appetite (Metabolism and nutrition disorders) | 1
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 1
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 1
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 1
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
bilateral leg cramping (Musculoskeletal and connective tissue disorders) | 1
finger stiffness (Musculoskeletal and connective tissue disorders) | 1
generalized body pain (Musculoskeletal and connective tissue disorders) | 1
hip pain (Musculoskeletal and connective tissue disorders) | 1
intermittent lower back pain (Musculoskeletal and connective tissue disorders) | 2
intermittent muscle cramps (hands) (Musculoskeletal and connective tissue disorders) | 1
posterior neck pain (Musculoskeletal and connective tissue disorders) | 1
twisted left ankle (Musculoskeletal and connective tissue disorders) | 1
10013573-Dizziness (Nervous system disorders) | 1
10013911-Dysgeusia (Nervous system disorders) | 3
10019211-Headache (Nervous system disorders) | 4
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 3
drowsiness (Nervous system disorders) | 1
10001497-Agitation (Psychiatric disorders) | 1
10002855-Anxiety (Psychiatric disorders) | 3
10012378-Depression (Psychiatric disorders) | 1
10038743-Restlessness (Psychiatric disorders) | 1
insomnia and nightmares (Psychiatric disorders) | 1
panic attacks (Psychiatric disorders) | 1
10006298-Breast pain (Reproductive system and breast disorders) | 4
10046904-Vaginal dryness (Reproductive system and breast disorders) | 1
10046912-Vaginal hemorrhage (Reproductive system and breast disorders) | 1
sensation in the R breast after the herceptin infusion (Reproductive system and breast disorders) | 1
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 3
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
10015090-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
10020201-Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
itchy throat (Respiratory, thoracic and mediastinal disorders) | 1
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 6
10037847-Rash acneiform (Skin and subcutaneous tissue disorders) | 2
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
10040865-Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
10054524-Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
acne (chin) (Skin and subcutaneous tissue disorders) | 1
hair follicle dicomfort (Skin and subcutaneous tissue disorders) | 1
mosquito bites (Skin and subcutaneous tissue disorders) | 1
pustules on face (Skin and subcutaneous tissue disorders) | 1
rash - arms and anterior chest (Skin and subcutaneous tissue disorders) | 1
skin changes R forarm (Skin and subcutaneous tissue disorders) | 1
10020407-Hot flashes (Vascular disorders) | 2
10020772-Hypertension (Vascular disorders) | 8
10021097-Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT02827877/Prot_SAP_000.pdf